CLINICAL TRIAL: NCT03456752
Title: The Impact of Perioperative Dexamethasone on Postoperative Outcome in Inflammatory Bowel Diseases.
Brief Title: Perioperative Dexamethasone on Postoperative Outcome in IBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEX-IBD
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases; Dexamethasone; Postoperative Ileus; Postoperative Complications
Keywords: Inflammatory Bowel Diseases; Glucocorticosteroids; Postoperative Outcome
MeSH Terms: conditions — Inflammatory Bowel Diseases; Postoperative Complications | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 8mg intravenously prior to anesthesia induction
  Interventions: Drug: Dexamethasone
- Control (Placebo Comparator): Normal Saline 1.6ml intravenously prior to anesthesia induction
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8mg intravenously prior to induction of anesthesia
  Arms: Dexamethasone
Drug: Normal saline — Normal saline 1.6ml intravenously prior to induction of anesthesia
  Arms: Control

SUMMARY:
The objective of this RCT is to determine the efficacy of a single preoperative dose of Dexamethasone for accelerating the recovery and reducing the incidence of postoperative complications in adult patients undergoing intestinal resection for inflammatory bowel disease.

DETAILED DESCRIPTION:
Patients undergoing surgery for IBD is associated with increased inflammatory response and incidence of prolonged ileus after surgery compared to other colorectal disease such as CRC. Previous studies have revealed that preoperative administration of glucocorticosteroids(GCs) decreased complications and length of postoperative length of hospital after major abdominal surgery as a likely consequence of attenuating the postsurgical inflammatory response. Also, a single dose of GCs did not increase complications in colorectal surgery. The aim of the study is to examine whether a single dose of dexamethasone prior to induction of anesthesia could promote the recovery of patients and reduce the incidence of prolonged ileus after surgery for IBD

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective open and laparoscopic small and large bowel operations for IBD, including Crohn's Disease(CD) and Ulcerative Colitis (UC).
2. ASA I-III

Exclusion Criteria:

1. Diabetes or hyperglycemia
2. Active gastric ulceration confirmed endoscopically
3. Presence of ongoing infection (such as IAS) or infective chronic diseases
4. Currently receiving systemic therapy with glucocorticoids with prednisolone >=20mg for over 6 weeks within 30 days prior to surgery.
5. Emergent surgery
6. Acute angle glaucoma
7. Pregnancy
8. Under 18 years of age
9. Known adverse reaction to dexamethasone
10. Extensive adhesiolysis
11. Carcinogenesis of intestinal tract

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Prolonged ileus | Day 30
  Prolonged POI was defined as if two or more of the following five criteria are met on day 4 postoperatively: nausea or vomiting; inability to tolerate an oral diet over last 24 h; absence of flatus over last 24 h; abdominal distension; and radiologic confirmation.

SECONDARY OUTCOMES:
PONV(Postoperative nausea and vomiting) and additional antiemetics given within 24hr after surgery | 24hr
  the incidence of any nausea, emetic episodes (retching or vomiting),or both (i.e., postoperative nausea and vomiting) during the first 24 postoperative hours.
Postoperative pain on POD 1, 3, and 5 | up to 1 week
  Visual analog scale (VAS) for pain description (0-10 visual analogue pain scale)
Postoperative fagitue score on POD 1, 3, and 5 | up to 1 week
  Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale (Version 4). The FACIT-IT score is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
GI-2 recovery | Day 30
  time to upper (first tolerance of solid food) and lower (first bowel movement) GI recovery (GI-2).
Blood WBC levels, preoperative and on postoperative 1,3 and 5 | Day 30
  Blood WBC levels, preoperative and on postoperative 1,3 and 5
Blood neutrophil percentage, preoperative and on postoperative 1,3 and 5 | Day 30
  Blood neutrophil percentage, preoperative and on postoperative 1,3 and 5
Serum C-reactive protein (CRP) level, preopperative and on postoperative 1,3 and 5 | Day 30
  Serum C-reactive protein (CRP) level, preopperative and on postoperative 1,3 and Serum C-reactive protein (CRP) level, preopperative and on postoperative 1,3 and Serum C-reactive protein (CRP) level, preopperative and on postoperative 1,3 and Serum C-reactive protein (CRP) level, preopperative and on postoperative 1,3 and
Serum Interleukin-6 (IL-6) level, preopperative and on postoperative 1,3 and 5 | Day 30
  Serum Interleukin-6 (IL-6) level, preopperative and on postoperative 1,3 and 5
Serum procalcitonin (PCT) level, preopperative and on postoperative 1,3 and 5 | Day 30
  Serum procalcitonin (PCT) level, preopperative and on postoperative 1,3 and 5
Body composition, preoperative and on POD 1 | Day 30
  body composition was determined using Bioelectrical impedance analysis (BIA)
Postoperative length of stay | Day 90
  in days
Postoperative morbidity | Day 30
  Documented using comprehensive complication index(CCI)
Postoperative surgical site infections (SSIs) | Day 30
  Including superficial SSIs and deep SSIs.
Overall cost of treatment | up to 1 year
  In Chinese Yuan (CNY)

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Gong, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang T, Xu Y, Yao Y, Jin L, Liu H, Zhou Y, Gu L, Ji Q, Zhu W, Gong J. Randomized Controlled Trial: Perioperative Dexamethasone Reduces Excessive Postoperative Inflammatory Response and Ileus After Surgery for Inflammatory Bowel Disease. Inflamm Bowel Dis. 2021 Oct 20;27(11):1756-1765. doi: 10.1093/ibd/izab065. PMID 33749741